CLINICAL TRIAL: NCT04979468
Title: Efficacy and Safety of Early Switching to Dolutegravir/Lamivudine (DTG/3TC) From INSTI-based Three-drug Regimens in HIV-1-infected Adults Previously naïve Who Achieve Virological Suppression
Brief Title: Early DOlutegravir/LAmivudine Switching After Virological Suppression (EDOLAS Study)
Acronym: EDOLAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa' Italiana Di Malattie Infettive E Tropicali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-004241-32
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Phase III, randomized, open-label, multicentre, active-controlled, non-inferiority study evaluating the efficacy and safety of early switching to dolutegravir/lamivudine (DTG/3TC) in single-pill, in HIV-1 infected individuals currently taking an INSTI-based three-drug first-line regimen for less than 18 months and who have been virologically suppressed with HIV-1 RNA <50 copies/mL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Other): Participants in Arm A will be randomized to switch to DTG/3TC 50/300 mg QD until week 48 (early switch).
  Interventions: Drug: DOVATO
- ARM B (Other): Participants in Arm B will continue the INSTI-based ART regimen until week 48, and then will be switched to DTG/3TC through week 96 (delayed switch).
  Interventions: Drug: DOVATO

INTERVENTIONS:
Drug: DOVATO — Dovato is a medicine for treating infection with human immunodeficiency virus type 1 (HIV-1), a virus that causes acquired immune deficiency syndrome (AIDS).
  Other Names: dolutegravir/lamivudine

SUMMARY:
Phase III, randomized, open-label, multicentre, active-controlled, non-inferiority study evaluating the efficacy and safety of early switching to dolutegravir/lamivudine (DTG/3TC) in single-pill, in HIV-1 infected individuals currently taking an INSTI-based three-drug first-line regimen for less than 18 months and who have been virologically suppressed with HIV-1 RNA <50 copies/mL

DETAILED DESCRIPTION:
The target population of this study is HIV-1-infected adults without previous virological failure, currently receiving any first-line, triple-drug ART having an INSTI (EVG/cobi, RAL QD, DTG, BIC) as anchor drug associated to any of the following dual NRTI backbone (ABC/3TC, TDF/FTC or TAF/FTC) with virological suppression (HIV-1 RNA < 50 copies/mL).

Participants will be randomly allocated 1:1 to switch to DTG/3TC 50/300 mg as a single pill qd until week 96 (Arm A, early switch) or to continue their INSTI-based ART triple regimen received at screening (Arm B, delayed switch) until week 52, when participants in Arm B with HIV-1 RNA< 50 cp/mL at week 48 will switch to DTG/3TC 50/300 mg qd as a single pill until week 100.

The drugs of both arms will be administered in an open-label manner throughout the entire duration of the study.

The primary analysis will take place after the last participant completes 52 weeks on therapy, to allow for the collection of a confirmatory viral load measurement in participants possibly presenting with HIV-1 RNA ≥50 cp/mL at the Week 48 visit.

If the second determination of HIV-1 RNA is <50 cp/mL, then the participant has not a virological rebound and will be considered eligible to switch to DTG/3TC at Week 52.

If the second determination of HIV-1 RNA is ≥50 cp/mL, then the participant will be considered protocol-defined virological failure, thus being ineligible to switch to DTG/ 3TC. These participants will be withdrawn from the study.

A preliminary interim analysis will be performed after 50% of the enrolled participants have reached the 24th week of study, always considering 4 weeks more (thus 28 weeks) to allow for the collection of a confirmatory viral load measurement in participants possibly presenting with HIV-1 RNA ≥50 copies/mL at Week 24.

At week 48, participants in Arm A (early switch) will continue DTG/3TC. At week 52, participants in Arm B (delayed switch) and with HIV-1 RNA < 50 copies/mL at week 48 will switch to DTG/3TC and will be followed until week 100.

The exploratory analyses at Week 96 will take place after the last participant completes 100 weeks on therapy, as needed, to allow for the collection of a confirmatory viral load measurement in participants presenting with HIV-1 RNA ≥50 copies/mL at Week 96.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 documented infection;
* Aged 18 years or older at the time of signing the informed consent;
* Stable INSTI-based first-line three-drug ART (switch between different NRTIs are allowed; e.g. from TDF/FTC to TAF/FTC or ABC/3TC, from TAF/FTC to TDF/FTC or ABC/3TC, from ABC/3TC to TAF/FTC or TDF/FTC). Any change of INSTI will not be allowed. Only the following regimens will be allowed:

  * RAL 1200 mg QD plus TDF/FTC or TAF/FTC;
  * RAL 1200 mg QD plus ABC/3TC;
  * EVG/COBI/FTC/TDF or EVG/COBI/FTC/TAF;
  * DTG plus TDF/FTC or TAF/FTC;
  * DTG/ABC/3TC or DTG plus ABC/3TC;
  * BIC/TAF/FTC
* Previous INSTI-based first-line ART lasting less than 18 months before screening;
* To have reached a HIV-1 RNA <50 copies/mL during INSTI first-line therapy for less than 12 months. At least a single HIV-1 RNA determination below the threshold within the 6 months before enrollment is required (if a following determination in present, this should not be ≥50 copies (cp)/mL)
* HIV-1 RNA below 50 copies/mL at the screening visit;
* No known allergy or intolerance to the study drugs or their components or drugs of their class;
* A female person is eligible to enter the study if it is confirmed that she is:

  * Not pregnant confirmed by a negative serum pregnancy test at both Screening and Day1;
  * Not breastfeeding;
  * Of non-childbearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy;
  * Of childbearing potential and agrees to utilize the protocol specified method of contraception (as defined in Appendix 1 -Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential) or be non-heterosexually active or practice sexual abstinence (defined as complete abstinence from penile-vaginal intercourse; periodic abstinence, e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) from screening throughout the duration of study treatment and for at least two weeks following discontinuation of study drugs;
* Being able to comply with the protocol requirements and restrictions;
* Signature of written Informed Consent Form (participants or legal guardian) before that any protocol-specified assessments are conducted.

Exclusion Criteria:

A person will be considered not eligible for inclusion in this study if any of the following criteria apply:

* Having failed virologically;
* Having changed the INSTI drug;
* Any major INSTI- or NRTI-resistance-associated mutation documented before starting ART;
* Women who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study;
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-Hbc), hepatitis B surface antigen antibody (anti-HBs) and, possibly, HBV DNA as follows:

  * Individuals positive for HBsAg are excluded;
  * Individuals negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded;
* HCV-RNA positivity needing for any hepatitis C virus (HCV) therapy during the study;
* Ongoing malignancy other than cutaneous Kaposi's sarcoma (not requiring systemic therapy), basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia;
* Active opportunistic infections requiring active treatment;
* Creatinine clearance of <50 mL/min/1.73m2 via CKD-EPI method;
* Individuals with severe hepatic impairment (Child Pugh class C) and/or unstable liver disease;
* Any verified Grade 4 laboratory abnormality at screening assessment;
* Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN) or ALT >3xULN and bilirubin >1.5xULN (with >35% direct bilirubin) at screening assessment;
* Receipt of investigational research agents within 30 days prior to study entry;
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening;
* Receipt of immunosuppressive medications or immune-modulators within the past 6 months;
* Individuals who in the investigator's judgment, poses a significant suicidality risk or with diagnosed major depression, Bipolar Disorders and Psychoses
* A life expectancy estimated as less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferior efficacy of switching | 48 weeks
  Proportion of participants with virological rebound (viral load ≥50 copies/mL or premature discontinuations, irrespective of reason, with last viral load ≥50 copies/mL) at week 48

SECONDARY OUTCOMES:
Efficacy of switching | 48 weeks
  Proportion of participants with HIV-1 RNA <50 copies/mL at week 48 (FDA Snapshot algorithm)
Safety and tolerability | 100 weeks
  Clinical and laboratory safety parameters; a descriptive analysis of all reported AEs and a quantitative analysis of AEs leading to treatment interruption/change will be used to evaluate long-term tolerability of the simplification treatment.
Immunologic response and dysfunction | 100 weeks
  Changes in CD4+ and CD8+ T-lymphocyte counts (absolute and percentage), and in CD4+/CD8+ ratio (as a measure of immune activation) in the peripheral blood from baseline to week 48 and 96.
Emergent drug resistance-associated mutations | 100 weeks
  Proportion of participants developing resistance-conferring mutations (to any drug class) by genotypic resistance test (GRT) in plasma or proviral DNA (in case of low viremia levels, <200 copies/mL) at protocol-defined virological failure (PDVF) will be cumulatively described throughout the study period.
RT and INSTI resistance-associated mutations | 100 weeks
  iral minority variants harboring resistance associated mutations (to any drug class) at the time of PDVF will be characterized in plasma or in proviral DNA (in case of low viremia levels, <200 copies/mL) by next generation sequencing. For the minority resistant variants detected (prevalence >1%), their resistance viral burden will be also evaluated.
Effects of the two strategies on Lipidic profile | 96 weeks
  Changes in fasting lipids (TC, LDL, HDL, non-HDL, TC/HDL) from baseline to w48 and 96.
Adherence levels to ARVs | 96 weeks
  Changes of self-reported adherence level and proportion of participants with different adherence level (95%; 90%; 80%) from baseline to week 48 and 96.
Evaluate neuropsychiatric symptoms. | 96 weeks
  Change in neuropsychiatric questionnaire scores, assessing mood, anxiety, sleep quality, and suicidality from baseline to week 24, 48 and 96.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Andreoni, P.I., Principal Investigator — Policlinico Universitario Tor Vergata; Alessandra Bandera, P.I., Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Alessandro Bartoloni, P.I., Principal Investigator — Azienda Ospedaliero-Universitaria Careggi; Stefano Bonora, P.I., Principal Investigator — Ospedale Amedeo di Savoia; Antonio Cascio, P.I., Principal Investigator — A.O.U. Policlinico "Paolo Giaccone"; Antonella Castagna, P.I., Principal Investigator — IRCCS Ospedale San Raffaele; Annamaria Cattelan, P.I., Principal Investigator — Azienda Ospedaliera di Padova; Roberto Cauda, P.I., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS; Benedetto Maurizio Celesia, P.I., Principal Investigator — ARNAS Garibaldi; Antonella d'Arminio Monforte, P.I., Principal Investigator — ASST Santi Paolo e Carlo - Presidio San Paolo; Antonio Di Biagio, P.I., Principal Investigator — Ospedale Policlinico San Martino di Genova; Massimo Antonio Di Pietro, P.I., Principal Investigator — Azienda Ospedaliero-Universitaria Careggi; Massimiliano Fabbiani, P.I., Principal Investigator — Azienda Ospedaliera Universitaria Senese; Roberto Gulminetti, P.I., Principal Investigator — Fondazione IRCCS Policlinico San Matteo; Giuseppe Lapadula, P.I., Principal Investigator — Ospedale San Gerardo di Monza; Giordano Madeddu, P.I., Principal Investigator — Strutture Ospedaliere - Cliniche San Pietro - AOU Sassari; Franco Maggiolo, P.I., Principal Investigator — ASST Papa Giovanni XXIII; Cristina Mussini, P.I., Principal Investigator — Azienda Ospedaliero-Universitaria di Modena; Massimo Puoti, P.I., Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda; Giuliano Rizzardini, P.I., Principal Investigator — ASST Fatebenefratelli Sacco; Stefano Rusconi, P.I., Principal Investigator — ASST Fatebenefratelli Sacco; Annalisa aracino, P.I., Principal Investigator — Azienda Ospedaliera Universitaria Policlinico di Bari; Laura Sighinolfi, P.I., Principal Investigator — Azienda Ospedaliera Universitaria Ferrara; Gabriella d'Ettorre, P.I., Principal Investigator — A.O.U. Policlinico Umberto I
Locations (23):
- Italy (23):
  - Azienda Ospedaliera Universitaria Policlinico di Bari, Bari, BA
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - ARNAS Garibaldi, Catania, CT
  - Azienda Ospedaliera Universitaria Ferrara, Ferrara, FE
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Ospedale Policlinico San Martino di Genova, Genova, GE
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI
  - IRCCS Ospedale San Raffaele, Milan, MI
  - ASST Fatebenefratelli Sacco, Milan, MI
  - ASST Santi Paolo e Carlo - Presidio San Paolo, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Ospedale San Gerardo di Monza, Monza, MI
  - Azienda Ospedaliera Universitaria di Modena, Modena, MO
  - A.O.U. Policlinico "Paolo Giaccone", Palermo, PA
  - Azienda Ospedaliera di Padova, Padua, PD
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Policlinico Universitario Tor Vergata, Roma, RM
  - Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS, Roma, RM
  - A.O.U. Policlinico Umberto I, Roma, RM
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM
  - Azienda Ospedaliera Universitaria Senese, Siena, SI
  - Strutture Ospedaliere - Cliniche San Pietro - AOU Sassari, Sassari, SS
  - Ospedale Amedeo di Savoia, Torino, TO

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: eCRF Home page — https://www.cr-technology.com/EDOLAS/